CLINICAL TRIAL: NCT06147167
Title: Effects of Individualized iTBS on Upper Limb Function After Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KYLL-202307-023
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-07

CONDITIONS: Upper Extremity Paresis; Stroke
Keywords: intermittent theta burst stimulation;; upper extremity paresis;; functional nearinfrared spectroscopy
MeSH Terms: conditions — Paresis; Stroke | interventions — Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- indvidualized iTBS (Experimental): In this arm of the study, participants undergo individualized intermittent theta burst stimulation (iTBS) subsequent to encephalography (EEG) testing. Three electrodes are strategically positioned on the first dorsal interosseous (FDI) hotspot to record the resting theta frequency, which is subsequently utilized as the theta frequency for theta burst stimulation (TBS). The participants receive this treatment regimen once daily, five times a week, over a total duration of three weeks.
  Interventions: Device: individualized intermittent theta burst sitmulation (iTBS)
- standard iTBS (Active Comparator): In this particular arm of the study, participants also undergo an initial electroencephalography (EEG) procedure. Subsequently, intermittent theta burst stimulation (iTBS) is administered using the standard theta burst stimulation frequency of 5Hz. The participants receive this treatment once daily, five times a week, over a total duration of three weeks.
  Interventions: Device: standard iTBS
- sham iTBS (Sham Comparator): In this arm, the treatment procedure is similar to the standard iTBS unless the coil is perpendicular to the scalp.
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: individualized intermittent theta burst sitmulation (iTBS) — Participants undergo daily sessions of individualized intermittent theta-burst stimulation (iTBS) administered with the MagStim stimulator (Rapid2, MagStim, Whiteland, United States). The intervention spans five days a week and extends over a three-week period. In this group, participants receive a personalized iTBS protocol comprising three pulses of stimulation delivered at 50 Hz, repeated every 200 ms. The stimulation frequency is tailored based on the electroencephalogram (EEG) results and is administered every 10 seconds, with a total duration of 190 seconds. The treatment is administered once a day for five days a week and continues for three weeks, with an immediate cessation in case of any discomfort. This study design ensures a meticulous and tailored approach to iTBS administration.
  Other Names: physical therapy; occupational therapy
  Arms: indvidualized iTBS
Device: standard iTBS — The MagStim stimulator (Rapid2, MagStim, Whiteland, United States) was employed in the current study. The intermittent theta-burst stimulation (iTBS) protocol utilized three pulses of stimulation delivered at a frequency of 50 Hz, with a repetition rate of every 200 ms. These pulses were organized into 2-second trains, repeated every 10 seconds, resulting in a cumulative duration of 190 seconds (equivalent to a total of 600 pulses). Notably, the administration of the treatment ceased promptly in the event of any participant discomfort.
  Other Names: physical therapy; occupational therapy
  Arms: standard iTBS
Device: sham stimulation — The device and protocol are identical to the standard iTBS, with the only difference being the orientation of the coil, which is perpendicular to the scalp.
  Other Names: physical therapy; occupational therapy
  Arms: sham iTBS

SUMMARY:
The primary objective of this clinical study is to assess the comparative efficacy of individualized intermittent theta burst stimulation (iTBS) in contrast to standard iTBS for individuals post-stroke experiencing upper limb impairment. The key inquiries addressed in this study encompass:

Enhancement of Upper Limb Function: The primary investigation seeks to determine whether individualized iTBS yields superior improvements in upper limb functionality compared to standard iTBS.

Long-Term Effects: This study endeavors to explore the sustained effects of both individualized and standard iTBS on upper limb function over an extended duration.

Neural Mechanisms Investigation: Functional near-infrared spectroscopy (fNIRS) will be employed to elucidate the neural mechanisms underlying the impact of iTBS on the enhancement of upper limb function.

Post-stroke individuals with upper limb impairment will undergo pre-treatment assessments, including motor function evaluations and fNIRS tests. Subsequently, they will be randomized into three groups: individualized iTBS, standard iTBS, and sham stimulation. Participants will undergo post-treatment assessments and follow-up evaluations.

The research team aims to discern disparities in the efficacy of different iTBS modalities. The central hypothesis posits that individualized iTBS will demonstrate superior efficacy in enhancing post-stroke upper limb function, with sustained effects persisting for a minimum of one month.

DETAILED DESCRIPTION:
This research constitutes a single-center, double-blind, randomized controlled study. Upon enrollment, baseline information is established through the assessment of upper limb function using the Fugl Meyer Assessment (FMA), the modified Rankin Scale, the Action Research Arm Test (ARAT), and a handgrip test. Additionally, functional near-infrared spectroscopy (fNIRS) is employed to assess brain function, providing insights into the patient's motor network.

Participants in the study are randomly assigned to one of three groups: individualized iTBS, standard iTBS, and sham stimulation. All participants undergo physical therapy and occupational therapy tailored to their functional evaluation. After three weeks of treatment, participants are required to complete the aforementioned assessments, with a follow-up evaluation scheduled one month post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. aging from 18-80
2. diagnosed as first-happened stroke,duration of the disease ranged from 1-3 months
3. upper extremity impairment
4. with mini-mental state examination>15
5. agree to participate in this study and sigh the informed consent

Exclusion Criteria:

1. with stroke history
2. have metal device within the body
3. with history of upper extremity trauma,fracture, and/or burn
4. serious conditions and can not finish the examination and treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-upper extremity | Befor and after the treatment, and 1 month after the treatment.
  Fugl-Meyer Assessment (FMA) scale is an index to assess the sensorimotor impairment in individuals who have had stroke. The FMA motor assessments for the upper fucntion with maximum score 66 points, including relflex activity, flexor synergy, extensor synergy, movement combining synergies, movement out of synergy,normal reflex, wrist function, hand function and coordination/speed, and sensory assessment.

SECONDARY OUTCOMES:
modified Rankin Scale | Befor and after the treatment, and 1 month after the treatment.
  The Modified Rankin Scale (mRS) assesses disability in patients who have suffered a stroke and is compared over time to check for recovery and degree of continued disability. A score of 0 is no disability, 5 is disability requiring constant care for all needs; 6 is death.
Action Research Arm Test | Befor and after the treatment, and 1 month after the treatment.
  The Action Research Arm Test (ARAT) is a 19 item observational measure used by physical therapists and other health care professionals to assess upper extremity performance (coordination, dexterity and functioning) in stroke recovery, brain injury and multiple sclerosis populations.Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally).
handrip test | Befor and after the treatment, and 1 month after the treatment.
  Hand grip test will be finished with a dynamometer.
functional nearinfrared spectroscopy | Befor and after the treatment, and 1 month after the treatment.
  The functional nearinfrared spectroscopy (fNIRS) is used to explore the motor network of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghui Wang, professor, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kong G, Wei L, Wang J, Zhu C, Tang Y. The therapeutic potential of personalized connectivity-guided transcranial magnetic stimulation target over group-average target for depression. Brain Stimul. 2022 Sep-Oct;15(5):1063-1064. doi: 10.1016/j.brs.2022.07.054. Epub 2022 Aug 2. No abstract available. PMID 35931377
- [Background] Klooster DCW, Ferguson MA, Boon PAJM, Baeken C. Personalizing Repetitive Transcranial Magnetic Stimulation Parameters for Depression Treatment Using Multimodal Neuroimaging. Biol Psychiatry Cogn Neurosci Neuroimaging. 2022 Jun;7(6):536-545. doi: 10.1016/j.bpsc.2021.11.004. Epub 2021 Nov 17. PMID 34800726
- [Background] Ferrarelli F, Phillips ML. Examining and Modulating Neural Circuits in Psychiatric Disorders With Transcranial Magnetic Stimulation and Electroencephalography: Present Practices and Future Developments. Am J Psychiatry. 2021 May 1;178(5):400-413. doi: 10.1176/appi.ajp.2020.20071050. Epub 2021 Mar 3. PMID 33653120
- [Background] Siddiqi SH, Trapp NT, Shahim P, Hacker CD, Laumann TO, Kandala S, Carter AR, Brody DL. Individualized Connectome-Targeted Transcranial Magnetic Stimulation for Neuropsychiatric Sequelae of Repetitive Traumatic Brain Injury in a Retired NFL Player. J Neuropsychiatry Clin Neurosci. 2019 Summer;31(3):254-263. doi: 10.1176/appi.neuropsych.18100230. Epub 2019 Apr 3. PMID 30945588
- [Background] Cassidy JM, Wodeyar A, Wu J, Kaur K, Masuda AK, Srinivasan R, Cramer SC. Low-Frequency Oscillations Are a Biomarker of Injury and Recovery After Stroke. Stroke. 2020 May;51(5):1442-1450. doi: 10.1161/STROKEAHA.120.028932. Epub 2020 Apr 17. PMID 32299324
- [Background] Cash RFH, Cocchi L, Anderson R, Rogachov A, Kucyi A, Barnett AJ, Zalesky A, Fitzgerald PB. A multivariate neuroimaging biomarker of individual outcome to transcranial magnetic stimulation in depression. Hum Brain Mapp. 2019 Nov 1;40(16):4618-4629. doi: 10.1002/hbm.24725. Epub 2019 Jul 22. PMID 31332903
- [Background] Ge R, Humaira A, Gregory E, Alamian G, MacMillan EL, Barlow L, Todd R, Nestor S, Frangou S, Vila-Rodriguez F. Predictive Value of Acute Neuroplastic Response to rTMS in Treatment Outcome in Depression: A Concurrent TMS-fMRI Trial. Am J Psychiatry. 2022 Jul;179(7):500-508. doi: 10.1176/appi.ajp.21050541. Epub 2022 May 18. PMID 35582784